CLINICAL TRIAL: NCT02574975
Title: Comparison of Different Methodologies Assessing Airway Responsiveness and Investigation of Treatment Efficacy of Budesonide /Formoterol in Asthmatics
Brief Title: Assessment of Airway Responsiveness and Treatment Efficacy in Asthmatics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ZhujiangH
Record Dates: First submitted 2015-10-08; First posted 2015-10-14 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Methacholine Chloride; Adenosine Monophosphate; Leukotriene D4; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Methacholine diagnosing group (Active Comparator): Methacholine bronchial provocation test was performed by using Jaeger spirometry with Aerosol Provocation System
  Interventions: Drug: methacholine
- Adenosine monophosphate diagnosing group (Experimental): Adenosine monophosphate bronchial provocation test was performed by using Jaeger spirometry with Aerosol Provocation System
  Interventions: Drug: adenosine monophosphate
- Leukotriene D4 diagnosing group (Experimental): Leukotriene D4 bronchial provocation test was performed by using Jaeger spirometry with Aerosol Provocation System
  Interventions: Drug: leukotriene D4
- Astograh diagnosing group (Experimental): Methacholine bronchial provocation test was performed by using Astograph Jupiter-21 airway reaction testing apparatus
  Interventions: Device: Astograph Jupiter-21 airway reaction testing apparatus
- budesonide /formoterol treatment group (Experimental): budesonide 160μg and formoterol 4.5ug,1 inhalation ,twice daily ,for three month
  Interventions: Drug: budesonide /formoterol

INTERVENTIONS:
Drug: methacholine — Methacholine,inhaled cumulative dosage 2.5mg
  Arms: Methacholine diagnosing group
Drug: adenosine monophosphate — Adenosine monophosphate ,inhaled cumulative dosage 40mg
  Arms: Adenosine monophosphate diagnosing group
Drug: leukotriene D4 — Leukotriene D4,inhaled cumulative dosage 2.4 μg
  Arms: Leukotriene D4 diagnosing group
Device: Astograph Jupiter-21 airway reaction testing apparatus — Methacholine bronchial provocation test was performed by using Astograph Jupiter-21 airway reaction testing apparatus
  Arms: Astograh diagnosing group
Drug: budesonide /formoterol — budesonide 160μg and formoterol 4.5ug,1 inhalation ,twice daily ,for three months in all participants (80 Anticipated)
  Other Names: Symbicort
  Arms: budesonide /formoterol treatment group

SUMMARY:
Bronchial asthma is a common chronic respiratory disease. Patients usually manifest variable symptoms (such as short of breath, chest tightness, cough, etc.) and variable airflow limitation and often associated with airway hyper-responsiveness and airway inflammation. About 1-18% of the global population suffered from the disease, causing huge economic burden for patients and countries. Airway reactivity measurement is an important way of diagnosis of asthma. Methacholine (Mch) bronchial provocation test(BPT) is the "gold standard" for the determination of airway reactivity, and other measuring methods(like adenosine monophosphate(AMP)-BPT, leukotriene D4(LTD4)-BPT, Astograph-BPT, etc.) were also brought into hot research fields. The investigators' purposes were to compare different kinds of methodologies(Mch,AMP,LTD4-BPT, Astograph-BPT) assessing airway responsiveness and to investigate treatment efficacy of budesonide /formoterol in asthmatics.

DETAILED DESCRIPTION:
This study composed of two parts, that were the diagnosing part and the treatment part.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed Asthmatic patients aged from14 to 65 years；
* Had a had a normal chest radiographic result；
* Had a baseline spirometry with the forced expiratory volume in one second (FEV1) of not less than 60% predicted；
* Without acute upper respiratory tract infection for the past 2 weeks

Exclusion Criteria:

* Smokers；
* Had a poor cooperation to the test or limited understandings;
* Had a past confirmed history of respiratory disease other than bronchial asthma (COPD, bronchiectasis, pulmonary thromboembolism, etc.) or other severe systemic disease（myocardial infarction, malignant tumor, etc.）;
* Pregnancy or breast-feeding women;
* Taken related drugs before measurements（Leukotriene receptor antagonists (LTRA) for 5 days，oral glucocorticosteroid or anti-histamine for 3 days，oral xanthenes or long-acting bronchodilators for 2 days，inhaled corticosteroid or long-acting bronchodilator for a day , short-acting bronchodilator for 4 hours ）

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
positive rate of BPT in each group | 3months
  comparing positive rates of BPT in experimental groups and control group

SECONDARY OUTCOMES:
Forced expiratory volume at one second（FEV1） | 3months
  change of FEV1 measured by pulmonary function test（PFT）at one month interval for 3 consecutive months
Fractional exhaled nitric oxide(FeNO) | 3months
  change of FeNO at one month interval for 3 consecutive months
Provocative dosage causing a 20% fall in FEV1(PD20-FEV1) | 3months
  change of PD20-FEV1 at one month interval for 3 consecutive months in each group

CONTACTS AND LOCATIONS:
Overall Officials: Huizhen Fan, Doctor, Study Chair — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China